CLINICAL TRIAL: NCT06861647
Title: iSITE: Investigation of Somatic Alterations in Tumours of the Eye
Acronym: iSITE
Status: Completed | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other); St. Bartholomew's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 242945
Record Dates: First submitted 2025-02-07; First posted 2025-03-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Somatic Mutation; Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Specimen Handling; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Uveal melanoma tissue samples from pathology archives and/or NHS REC approved research tissue banks. Eye tumour tissue biopsies, surgical waste material from eye tumour operations, vitreous fluid and blood samples. Healthy eye, blood and liver samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- A (Primary uveal melanoma): Prospective collection, primary uveal melanoma. If patients have previously collected samples, consent will be requested to also obtain these samples.
  Interventions: Other: sample collection; Other: Discussing study/seeking consent; Other: Completion of Study Questionnaire; Other: Blood Sample
- B1 (Metastatic uveal melanoma): Prospective collection, metastatic uveal melanoma. If patients have previously collected samples, consent will be requested to also obtain these samples.
  Interventions: Other: sample collection; Other: Discussing study/seeking consent; Other: Completion of Study Questionnaire; Other: Blood Sample
- B2 (Metastatic uveal melanoma, precollected only): Previously collected and stored tissue samples, retrospective collection only, metastatic uveal melanoma
- C (Conjunctival melanoma): Previously collected and stored tissue samples, retrospective collection only, metastatic conjunctival melanoma ,

INTERVENTIONS:
Other: sample collection — sample collection of surplus samples not needed for diagnostic or pathological requirements
  Groups: A (Primary uveal melanoma); B1 (Metastatic uveal melanoma)
Other: Discussing study/seeking consent — An NHS or CRN staff member will inform patients of the nature and objectives of the study, go through the participant information sheet, highlighting possible risks associated with their participation and reiterate the voluntary nature of this study. Patients will be given opportunities to ask questions pertaining to the study. If the potential participant is still interested in taking part, written informed consent for the study will then be received and a copy of the informed consent will be given to the participant to keep.
  Groups: A (Primary uveal melanoma); B1 (Metastatic uveal melanoma)
Other: Completion of Study Questionnaire — Patient will complete in own time. To take place in a routine outpatient clinic appointment
  Groups: A (Primary uveal melanoma); B1 (Metastatic uveal melanoma)
Other: Blood Sample — To take place in an outpatient clinic.
  Groups: A (Primary uveal melanoma); B1 (Metastatic uveal melanoma)

SUMMARY:
Modern DNA sequencing technologies enable researchers to identify mutations that have been acquired during the lifetime of patients (somatic mutations). Some of these somatic mutations occur in cancer genes and increase the risk of developing cancer. This study will apply such sequencing technologies to cancers of the eye (ocular melanoma) in order to identify mutations associated with these cancers. Sequencing patients at different stages of their disease will allows us to build a timeline of the order of mutations that occur at each stage. This information can be used to understand how these cancers develop, spread (metastasise) and respond to treatment. Furthermore, the study will look at which of these somatic mutations are present in the blood, by collecting blood samples and sequencing fragments of DNA which have been released by tumours into the bloodstream (circulating tumour DNA, ctDNA). This will determine whether ctDNA can be used as a way of monitoring mutations present in the tumour. This study will provide much needed insight into a rare and understudied cancer type, with the long-term aim of improving the survival of patients by identifying key mutations to develop novel therapies against.

DETAILED DESCRIPTION:
Uveal melanomas are rare cancers that arise from pigment cells (melanocytes) in the eye. Like most rare cancers, limited interest in developing new therapies and a lack of clinical trials contributes towards relatively worse survival rates compared with common cancers. Following treatment of uveal melanoma with either surgical removal of the eye (enucleation) or local radiation (plaque brachytherapy), approximately half of all patients will develop metastases (new tumours). Most patients will die within a few months despite current therapies.

Conjunctival melanomas (cancer of the surface of the eye which lines the inside of the eyelids) are an extremely rare subset of eye cancers which also have poor survival outcomes once metastasised. Modern DNA sequencing technologies enable researchers to identify mutations acquired during the lifetime of an individual (these are known as somatic mutations). Some of these somatic mutations occur in cancer-associated genes, and increase the risk of developing cancer. This study will use sequencing technologies to look to identify mutations associated with cancers of the eye. By sequencing at different stages of the disease we hope to build a timeline of the order of mutations that occur during eye cancer development. The investigators will also generate cell line models to try and understand how these cancers develop, spread (metastasise) and respond to treatments. The investigators will also look at which somatic mutations are detectable in blood. Blood samples will be collected regularly from participants and circulating tumour DNA, (ctDNA, fragments of DNA released by tumours into the bloodstream) will be sequenced. The investigators will determine whether the mutations present in ctDNA can be used as an indicator of disease progression.

This study will provide much needed insight into a rare and understudied cancer type, with the aim of improving the survival of patients by identifying key mutations to develop novel therapies against.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age or over
* Histological diagnosis of primary or recurrent/metastatic ocular melanoma*.
* Healthy eye, blood and liver samples stored in biobanks with consent for use in research.

  * *With the exception of primary uveal melanoma where a clinical diagnosis is sufficient. A diagnostic accuracy of >99% is achieved using the combination of ophthalmoscopy (examination of the back of the eye), fundus photography (photograph of the back of the eye) and an eye ultrasound.

Exclusion Criteria:

* Patients < 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research study will include participants with primary uveal melanoma and/or metastatic uveal melanoma and participants with conjunctival melanoma.
  A member of the participant's clinical care team, a research nurse or member of the Clinical Research Network (CRN) will have access to patient records to identify potential participants and check whether they meet the eligibility criteria and if there are previously collected available samples.
  Patients who have, and those who have not, previously given written consent for their samples that were obtained during standard procedures of treatment, to be used in research, will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Measuring what somatic mutations are acquired during development and metastases in uveal melanomas and conjunctival melanomas. | 6.5 years
  Tracking the mutational changes of a tumour in the same patient over time will allow the investigators to determine the order in which mutations are acquired and therefore provide insight into their roles in disease biology. Most studies have sequenced primary tumours and metastatic tumours from different patients. This makes comparison between the two groups of tumours difficult due to the presence of mutations specific to patients, but not necessarily important for cancer development. To determine the relevance of these commonly altered genes, a larger number of paired tumours will be sequenced.
Measure whether tumour intratumoural heterogeneity (the mixture of different tumour cell types within one tumour) is associated with a poor clinical outcome. | 6.5 years
  There is emerging evidence that diverse populations of cells exist in different regions within a single tumour (intratumoural heterogeneity) in uveal melanoma. This is a result of the development of different groups of mutations (subclones) which evolve - a reflection of the adaptive nature of cancer over time. Intratumoural heterogeneity has been linked with poor clinical outcomes in other cancer types. This study will determine what subclones exist, and to what extent they are associated with poor clinical outcomes in uveal and conjunctival melanoma.
  Samples at different time points from the same patient, and samples across different regions within the same tumour, will undergo sequencing of the whole genome, whole exome or targeted sets of cancer genes. This will allow identification of somatic alterations from base substitutions to larger genome rearrangements, and comparisons to be made between the burden and type of somatic alternations identified.
Measuring the burden and prevalence of somatic mutations in normal and cancer samples of tumours of the eye | 6.5 years
  Samples at different time points from the same patient, and samples across different regions within the same tumour, will undergo sequencing of the whole genome, whole exome or targeted sets of cancer genes. This will allow identification of somatic alterations from base substitutions to larger genome rearrangements, and comparisons to be made between the burden and type of somatic alterations identified.

SECONDARY OUTCOMES:
Do mutations detected in circulating tumour DNA reflect the somatic mutations found within the tumour and the effectiveness of this measure as a means of monitoring tumour evolution, and disease progression. | 6.5 years
  Cohorts A and B1: Uveal melanoma only.
  This study will include longitudinal blood sampling for the detection of mutations in ctDNA. If these mutations are found to be a real-time reflection of the mutations present within the tumour, this would be a valuable minimally-invasive approach to studying tumour evolution and monitoring disease.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Ying Chan, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom